CLINICAL TRIAL: NCT00051818
Title: Immune and Viral Outcomes of HIV-1 Therapy Interruption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Wistar Institute (Other)
Responsible Party: Principal Investigator, Luis Montaner, Professor and Director, HIV-1 Immunopathogenesis Laboratory, The Wistar Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01AI048398-01 (NIH); AI048398
Record Dates: First submitted 2003-01-16; First posted 2003-01-24 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2005-12

CONDITIONS: HIV Infections
Keywords: chronic HIV infection; treatment interruption; HIV-specific immune response; immune response; virological response; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Treatment interruption/reinitiation schedule

SUMMARY:
The purpose of this study is to determine if stopping anti-HIV drugs for a period of time is safe and effective for enhancing the immune function of patients with HIV.

DETAILED DESCRIPTION:
Our preliminary studies have shown that structured treatment interruption of highly active antiretroviral therapy (HAART) may boost patients' immune responses to HIV-1. In this study, we will test the hypothesis that repeated structured treatment interruptions will increase HIV-1 immunity and result in better control of viral replication than in controls. We will test this hypothesis by determining time to viral rebound after withdrawal of antiretroviral therapy in a randomized, non-blinded study of a well-characterized subject population from a single center. Patients in this study will be randomized to either treatment interruption or control groups. Patients will be monitored for adherence to therapy and changes in immune status following HAART interruption. CD4 percentage, CD 4 and CD8 mediated anti-HIV-1 responses, cell surface T-cell antigen expression, and thymic function will be assessed.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 positive
* HIV RNA < 500 copies/ml on a regimen of two nucleoside reverse transcriptase inhibitors (NRTIs) and either one protease inhibitor (PI) or one nonnucleoside reverse transcriptase inhibitor (NNRTI) for 6 months prior to study entry - HIV RNA < 50 copies/ml at study screening
* CD4 > 400 cells/mm3 with CD4 nadir of > 100 cells/mm3
* Agree to Medication Event Monitoring System monitoring of one component of antiretroviral regimen
* HIV-1 viral load >10,000 copies/ml at any time prior to initiating the current uninterrupted HAART regimen
* Willing to abstain from all immunomodulatory drugs during the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-09; Primary Completion 2003-05 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Viral suppression in the absence of therapy, compared to a structured treatment interruption (STI) group maintaining continual suppression

SECONDARY OUTCOMES:
Safety of sequential STIs
changes in immune reconstitution in relation to sequential STIs, including CD4 T-cell changes, recall responses, and T-cell activation, as measured by cell surface antigen changes
genotypic changes occurring in HIV-1 protease and reverse transcriptase regions after sequential STIs and their relation to clinical failure under the ART regimen at study entry

CONTACTS AND LOCATIONS:
Overall Officials: Luis J. Montaner, Principal Investigator — The Wistar Institute
Locations (1):
- The Wistar Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Montaner LJ. Structured treatment interruptions to control HIV-1 and limit drug exposure. Trends Immunol. 2001 Feb;22(2):92-6. doi: 10.1016/s1471-4906(00)01809-3. PMID 11286710
- [Result] Papasavvas E, Kostman JR, Mounzer K, Grant RM, Gross R, Gallo C, Azzoni L, Foulkes A, Thiel B, Pistilli M, Mackiewicz A, Shull J, Montaner LJ. Randomized, controlled trial of therapy interruption in chronic HIV-1 infection. PLoS Med. 2004 Dec;1(3):e64. doi: 10.1371/journal.pmed.0010064. Epub 2004 Dec 28. PMID 15630469
- [Result] Papasavvas E, Grant RM, Sun J, Mackiewicz A, Pistilli M, Gallo C, Kostman JR, Mounzer K, Shull J, Montaner LJ. Lack of persistent drug-resistant mutations evaluated within and between treatment interruptions in chronically HIV-1-infected patients. AIDS. 2003 Nov 7;17(16):2337-43. doi: 10.1097/00002030-200311070-00008. PMID 14571185
- [Derived] Papasavvas E, Azzoni L, Ross BN, Fair M, Howell BJ, Hazuda DJ, Mounzer K, Kostman JR, Tebas P, Montaner LJ. Comparable HIV suppression by pegylated-IFN-alpha2a or pegylated-IFN-alpha2b during a 4-week analytical treatment interruption. AIDS. 2021 Oct 1;35(12):2051-2054. doi: 10.1097/QAD.0000000000002961. PMID 34049356